CLINICAL TRIAL: NCT04186286
Title: A Randomized Crossover Study of Propranolol Versus Ivabradine in Postural Tachycardia Syndrome (POTS)
Brief Title: Crossover Study of Propranolol vs Ivabradine in POTS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Dysautonomia International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB19-1437
Record Dates: First submitted 2019-11-21; First posted 2019-12-04 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Postural Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Ivabradine; Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 1st drug Ivabradine (Active Comparator): Patients will take Ivabradine first followed by Propranolol and Placebo
  Interventions: Drug: Ivabradine 4-week course; Drug: Propranolol 4-week course; Drug: Placebo 4-week course
- 2nd drug Ivabradine (Active Comparator): Patients will take either Propranolol or placebo first and then Ivabradine
  Interventions: Drug: Ivabradine 4-week course; Drug: Propranolol 4-week course; Drug: Placebo 4-week course
- 3rd drug Ivabradine (Active Comparator): Patients will take Propranolol and placebo first and then Ivabradine
  Interventions: Drug: Ivabradine 4-week course; Drug: Propranolol 4-week course; Drug: Placebo 4-week course

INTERVENTIONS:
Drug: Ivabradine 4-week course — After a baseline screening assessment following a washout period of 7 days, participants will be randomized to start with a 4-week course of ivabradine.
  Other Names: Lancora
Drug: Propranolol 4-week course — After a baseline screening assessment following a washout period of 7 days, participants will be randomized to start with a 4-week course of propranolol.
  Other Names: Inderal
Drug: Placebo 4-week course — After a baseline screening assessment following a washout period of 7 days, participants will be randomized to start with a 4-week course of placebo

SUMMARY:
1.0 BACKGROUND Postural tachycardia syndrome (POTS) is a disorder of chronic orthostatic intolerance characterized by symptoms of palpitations, lightheadedness, chest discomfort, shortness of breath, blurred vision, and mental clouding. These symptoms occur during standing and are associated with a marked increase in heart rate (HR) in the absence of hypotension, which typically resolve when sitting or lying down. Most importantly, POTS is associated with a very poor quality of life and significant functional disability. POTS patients commonly experience mental clouding ("brain fog") even while lying down or seated, which poses significant limitations to daily activities .

Unfortunately, there is a relative paucity in the literature assessing therapies for POTS patients. Given that excessive tachycardia on standing is a fundamental component of this syndrome, a handful of studies have evaluated medications that reduce HR. Ivabradine is newer drug that is a selective If channel blocker that reduces HR without affecting other cardiovascular functions.

2.0 RATIONALE / STUDY PURPOSE The investigators propose to compare the efficacy of propranolol and ivabradine on HR response to standing, and symptom burden in patients with POTS.

3.0 Study Design This will be a single-center double-blind placebo-controlled randomized crossover trial conducted in patients with POTS to compare effects of (1) oral ivabradine 5 mg bid plus placebo BID (to fill out a QID schedule); (2) oral propranolol 10 mg qid; and (3) oral placebo qid in POTS patients. After a baseline screening assessment following a washout period of 7 days, participants will be randomized to start with a 4-week course of either ivabradine, propranolol or placebo. The other two treatments will be given in separate 4-week courses with a 7-day washout period between phases, with each participant acting as his or her own control. At the end of each 4-week phase, participants will complete the symptom-rating and HRQOL questionnaires, and also undergo tilt table testing to assess the change in HR at 10 min with head up tilt.

Participants will undergo POTS testing at baseline and at the end of each 4-week treatment course. This will involve a total of 4 separate study visits.

DETAILED DESCRIPTION:
1.0 BACKGROUND Postural tachycardia syndrome (POTS) is a disorder of chronic orthostatic intolerance characterized by symptoms of palpitations, lightheadedness, chest discomfort, shortness of breath, blurred vision, and mental clouding. These symptoms occur during standing and are associated with a marked increase in heart rate (HR) in the absence of hypotension, which typically resolve when sitting or lying down. Most importantly, POTS is associated with a very poor quality of life and significant functional disability. POTS patients commonly experience mental clouding ("brain fog") even while lying down or seated, which poses significant limitations to daily activities .

Unfortunately, there is a relative paucity in the literature assessing therapies for POTS patients. Given that excessive tachycardia on standing is a fundamental component of this syndrome, a handful of studies have evaluated medications that reduce HR. In a randomized crossover study of 54 patients with POTS, low-dose propranolol (10-20 mg PO) was found to acutely reduce standing HR compared to placebo. Further, there was greater improvement in symptom burden (quantified using the Vanderbilt Orthostatic Symptom Score [VOSS]) from baseline to 2 hours in patients treated with propranolol compared to placebo.

Ivabradine is newer drug that is a selective If channel blocker that reduces HR without affecting other cardiovascular functions. In non-randomized reports, it has been shown to improve symptoms in patients with POTS. In a case series of 22 patients, approximately 60% of patients with POTS treated with ivabradine had symptom improvement

2.0 RATIONALE / STUDY PURPOSE Patients with POTS suffer great disability and currently used pharmacologic therapies require more rigorous study. Currently, there are no studies comparing the relative efficacy of propranolol and ivabradine in patients with POTS.

We propose to compare the efficacy of propranolol and ivabradine on HR response to standing, and symptom burden in patients with POTS. This would be the first study to compare the relative efficacy of ivabradine to propranolol in POTS. The results of this exploratory study may help inform design of a larger multicenter clinical trial investigating the use of ivabradine or propranolol in POTS over time. We will test the null hypothesis that the heart rate lowering response to ivabradine is not different than the heart lowering response of propranolol.

In addition, we propose to assess sleep complaints and sleep quality using questionnaire and actigraphy based assessments.

3.0 Study Design This will be a multi-center double-blind placebo-controlled randomized crossover trial conducted in patients with POTS to compare effects of (1) oral ivabradine 5 mg bid plus placebo BID (to fill out a QID schedule); (2) oral propranolol 10 mg qid; and (3) oral placebo qid in POTS patients. After a baseline screening assessment following a washout period of 7 days, participants will be randomized to start with a 4-week course of either ivabradine, propranolol or placebo. The other two treatments will be given in separate 4-week courses with a 7-day washout period between phases, with each participant acting as his or her own control. At the end of each 4-week phase, participants will complete the symptom-rating and HRQOL questionnaires, and also undergo tilt table testing to assess the change in HR at 10 min with head up tilt.

Participants will undergo POTS testing at baseline and at the end of each 4-week treatment course in the Libin Cardiovascular Institute TRW Human Physiology Research space. This will involve a total of 4 separate study visits.

•• Studies will start between 8-9am, with the patient in a fasting state (to avoid acute hemodynamic effects from eating).

* Prior to hemodynamic data collection, a brief medical history will be conducted to ensure that the medications have not changed, and that there are not new medical issues that would make the study unsafe or imprudent.
* Participants will be instrumented for continuous beat-to-beat BP and electrocardiographic monitoring. BP will be monitored continuously using a finger volume clamp method (Nexfin, BMEYE Inc.) and calibrated with intermittent brachial cuff measurements using a standard automatic BP monitor (IVY Model 450C, IVY Medical, Branford, CT, USA) or by using Finapres NOVA, Finapres Medical Systems .
* Baseline seated continuous data (EKG signals and continuous BP will be collected for ~10 min).
* Neuropsychological testing of the cognitive domains of memory, attention and executive function will be assessed using the Cambridge Neuropsychological Test Automated Battery (CANTAB) while seated.
* The patient will be asked to stand and repeat portions of the CANTAB tests
* Baseline lying down continuous data (EKG signals and continuous BP will be collected for ~10 min).
* The patient will then be strapped onto the tilt table and then tilted to 80° head-up for 10 minutes with continuous hemodynamic data collection. Oxygen saturation will be assessed from a finger probe. End-tidal CO2 will be measured using nasal prongs.
* Participants will be asked to comment on any side effects or unrated symptoms.
* VOSS ratings will be collected at the end of tilt.
* Participants and the research staff will be asked to "guess" at which intervention was given on that study day (not applicable to baseline visit).
* After the study is finished, we will remove the recording patches, and electrodes. This testing day will last about 3 hours.

Upon conclusion of the tilt testing, we will connect patients to a 24-hour Holter monitor for continuous ECG and HR monitoring. Participants will return the monitoring device the following day.

This testing protocol will be repeated at baseline, and at the end of phase 1, 2, and 3 with different study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Postural Tachycardia Syndrome
* Age between 18-60 years
* Men and women are eligible
* Able and willing to provide informed consent

Exclusion Criteria:

* Seated resting heart rate < 70 bpm in the absence of rate-lowering medications
* Supine blood pressure < 90/60 mmHg
* Overt cause for postural tachycardia, i.e., acute dehydration, prolonged bed rest
* Presence of underlying structural heart disease including:
* Valvular disease (i.e. moderate or greater valvular stenosis or regurgitation)
* History of heart failure
* Greater than mild left ventricular systolic impairment
* Hypertrophic cardiomyopathy
* Known coronary artery disease or prior myocardial infarction
* History of tachyarrhythmias including:
* Supraventricular tachycardia, atrial tachycardia, atrial fibrillation / flutter
* Ventricular tachyarrhythmias
* Pre-existing long QT interval (e.g. known congenital long QT syndrome, or QT interval >500 ms)
* History of sick sinus syndrome or high degree AV block
* Presence of a pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy device
* Diabetes mellitus or history of hypoglycemic episodes
* History of bronchospasm or uncontrolled asthma
* Pregnant (by history or serum test) or breast-feeding
* Inability to safely withdraw from existing beta-blockers or ivabradine prior to the study day
* Concomitant use of class I and III antiarrhythmic agents, or non-dihydropyridine calcium channel blockers
* Concomitant use of strong cytochrome P450 3A4 (CYP 3A4) inhibitors
* Severe hepatic impairment
* Any contraindication to propranolol or ivabradine not specifically listed above as per the product monographs.
* Unable to give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HR | 4 weeks
  the ∆HR from supine to standing on head-up tilt at 10 minutes after the 4 weeks each of patient taking Ivabradine, Propranolol and Placebo

SECONDARY OUTCOMES:
Vanderbilt Orthostatic Symptoms Score | 4 weeks
  change in symptom burden quantified by the VOSS at 10 minutes of head-up tilt after the 4 weeks each of patient taking Ivabradine, Propranolol and Placebo

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada